CLINICAL TRIAL: NCT05221333
Title: Assessment of Safety and Performance of an Investigational Wearable Injector in Healthy Volunteers
Brief Title: Sorrel 25R Injector - Sorrel Clinical Study Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eitan Medical (Industry)
Collaborators: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: VAL-15144-0005662
Record Dates: First submitted 2021-08-19; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2021-08

CONDITIONS: Injection Site; Injection Site Reaction; Injection Site Irritation
Keywords: wearable injector
MeSH Terms: conditions — Injection Site Reaction

STUDY DESIGN:
Intervention Model Description: a single group of health participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Healthy participants (Other): Up to 25ml of saline administered through OBI
  Interventions: Device: Sorrel Wearable Injector

INTERVENTIONS:
Device: Sorrel Wearable Injector — Use of Sorrel Wearable Injector in pilot study

SUMMARY:
A prospective, open-label, single-center pilot study to evaluate the performance, safety and usability of the investigational SWI Device in healthy volunteers.

DETAILED DESCRIPTION:
A prospective, open-label, single-center pilot study to evaluate the performance, safety and usability of the investigational SWI Device in healthy volunteers.

The study will enroll up to 25 healthy adult subjects. Each subject will perform a maximum of 5 visits during the study over a period of approximately 2 months; a virtual visit for informed consent, two in-person visits for device evaluation, and two follow-up virtual visits to evaluate the skin and surrounding tissue for adverse events.

ELIGIBILITY:
Inclusion Criteria:

Age 18 to ≤ 40 years.

Subject understands the English language, understands the risks, benefits, and alternatives to this research study, and is willing and able to give written informed consent.

Subject has no active signs/symptoms of a viral infection for 10 days prior to visit # 2.

Body Mass Index between 20 to 35 kg/m2 (inclusive).

Subject willing and able to comply with study procedures.

American Society of Anaesthesiology Physical status (ASA PS) classification 1

Exclusion Criteria:

Current use of aspirin at a daily dose > 81 mg,

Current use of any medication that may adversely affect blood coagulation (i.e. warfarin, Xarelto, Eliquis etc.)

Presence of any tattoos, discoloration, acne, scars, bruises, cuts, abrasions, rashes, hernias, or inflammation within the skin or subcutaneous tissue of the abdomen that could interfere with the infusion of saline or observation of study results, at the discretion of the investigator..

History of significant skin allergy, irritation, or hypersensitivity to medical adhesives or adhesive tape.

History of significant allergic reaction to medical saline solution.

History of significant allergic reaction to the skin antiseptic solutions alcohol or chlorhexidine.

History of any neurologic disease that may affect the perception of pain/discomfort (stroke, peripheral neuropathy).

Current use of any medication that may affect the perception of pain/discomfort (opioids, NSAIDs, topical local anesthetics) at the discretion of the investigator.

Current use of any medical condition or medication that to the opinion of the investigator may affect the risk for a serious adverse event

Female of childbearing age with a positive pregnant test, or currently breast feeding.

Study subject refuses to allow clipping of excess abdominal hair at the site of device placement

Any current or unstable cardiac, pulmonary, hepatic, renal, neurologic, gastrointestinal, endocrine, immune, endocrine, musculoskeletal, coagulation disorder, or infectious disease which in the opinion of the Investigator would place the subject at risk or influence the conduct of the study, or interpretation of the results.

Current participation in another clinical drug or device study.

Inability of the subject to comply with all study procedures.

Inability of the subject to understand the information required for monitoring their infusion sites.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Reliability of SWI | 24 hours
  70% successful injection confirmed by visual inspection of investigator

SECONDARY OUTCOMES:
Incidences of Treatment Emergent Adverse Events of SWI | 1 month
  Evaluation of AEs
Pain associated with use of SWI | 1 month
  Pain assessment based on visual analog scale (VAS), higher score means worse outcome

OTHER OUTCOMES:
Overall experience of SWI | 24 hours
  Assessment of overall experience based on patient questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Marc C Torjman, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot study for internal use only